CLINICAL TRIAL: NCT06864091
Title: Esthetic Evaluation of Facial Prostheses Fabricated Using Direct and Indirect Additive Manufacturing Techniques: A Pilot Randomized Crossover Clinical Trial
Brief Title: Different Manufacturing Techniques of Facial Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatima Elmougi, Doctor, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1024
Record Dates: First submitted 2025-02-27; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Facial Defects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Mould Making (Experimental)
  Interventions: Other: Direct Mould Making
- Indirect Mould Making (Experimental)
  Interventions: Other: Indirect Mould Making
- Rapid Manufacturing (Experimental)
  Interventions: Other: Rapid Manufacturing

INTERVENTIONS:
Other: Rapid Manufacturing — The first intervention (I1) involves direct printing of the final prosthesis (rapid manufacturing, RM). The final prosthesis will be printed using a biocompatible rubber-like printable soft resin (Biomed Flex 80A resin, Formlabs, USA), and then will be colored and characterized to match the surrounding anatomy.
  Arms: Rapid Manufacturing
Other: Direct Mould Making — In the second intervention (I2), the negative mold will be achieved directly, will be virtually designed based on an inverted STL file of prosthesis prototype/ pattern (direct mold making, DMM).
  Arms: Direct Mould Making
Other: Indirect Mould Making — the negative mold will be fabricated indirectly by printing the prosthesis prototype from resin for subsequent mold fabrication (indirect mold making, IMM). The printed prototype will be tried on the patient and adjusted in terms of shape, size and marginal fit.
  After the try-in stage the prototype will be duplicated into wax by using silicone rubber molding and a conventional stone mold will be fabricated.
  Arms: Indirect Mould Making

SUMMARY:
All participants will undergo 3-dimentional facial scan and the defect site will be scanned using intraoral scanner. the data will be extracted in Standard tessellation Language (STL) and used in virtual prosthesis reconstruction.

* (Group 1) involves direct printing of the final prosthesis using biocompatible rubber-like printable soft resin.
* Group 2, involves direct manufacturing of the negative mold, it will be virtually designed based on an inverted STL file of prosthesis prototype/ pattern.
* Group 3, involves fabrication of the negative mold indirectly by printing the prosthesis prototype from resin and then duplicating it into wax and a conventional stone mold will be fabricated.
* The negative molds of both groups 2&3 will be used in packing medical grade silicone (to cast the final prosthesis.
* All final prostheses will be colored and characterized to match the surrounding anatomy.
* Esthetic outcomes will be assessed using VAS scale by answering operator and patient related questionnaires. The patient related questionnaire will be translated to the patients and responses will be recorded. For each patient, a score will be given from 1-5.
* Prosthesis accuracy will be assessed using Medit software, comparing the scan of the final prosthesis to the STL of the prosthesis design and the root mean square (RMS) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cartilaginous facial defects, i.e: auricular and nasal defects.
2. Patients between 20-60 years old.
3. Post traumatic patients with facial defects.
4. Patients with congenital facial defects.
5. Patients with failed facial surgical construction.
6. Compliant and cooperative patients.

Exclusion Criteria:

1 - Patients having risk of tumor recurrence in the defect area. 2- Patients undergoing radiotherapy or chemotherapy treatment. 3- Patients with any debilitating disease. 4- Patients with any type of psychosomatic disorder. 5- Patients with allergy to any of the materials used.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Esthetic Outcomes | 3 months
  Esthetic outcomes will be assessed using VAS scale by answering operator and patient related questionnaires. The patient related questionnaire will be translated to the patients and responses will be recorded. For each patient, a score will be given from 1-5.

SECONDARY OUTCOMES:
Prosthesis Accuracy | 3 months
  Prosthesis accuracy will be assessed using Medit software, comparing the scan of the final prosthesis to the STL of the prosthesis design and the root mean square (RMS) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No